CLINICAL TRIAL: NCT04629001
Title: Effect of Covid-19 on Outcomes of Pregnancy
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Armia Michael, Physician, Assiut University
Other Study IDs: 12789
Record Dates: First submitted 2020-11-12; First posted 2020-11-16 (Actual); Last update posted 2020-11-16 (Actual); Status verified 2020-11

CONDITIONS: Pregnancy Without Complications Except Getting Covid-19 Infection
Keywords: pregnancy; Covid-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- with Covid-19 infection
  Interventions: Diagnostic Test: Covid-19 PCR , IGM
- without Covid-19 infection
  Interventions: Diagnostic Test: Covid-19 PCR , IGM

INTERVENTIONS:
Diagnostic Test: Covid-19 PCR , IGM — test for Covid-19

SUMMARY:
To study the effect of getting Covid-19 infection during pregnancy on the outcomes of the mother and the fetus including morbidity and mortality

ELIGIBILITY:
Inclusion Criteria:

* Normal single pregnancy

Exclusion Criteria:

* Pregnancy with any chronic diseases
* Multiple pregnancy

Ages: 18 Years to 40 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes
Study Population: Female in Reproduction age
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-09-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Fetal morbidity | 28 days

CONTACTS AND LOCATIONS:
Locations (1):
- Medicine, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided